CLINICAL TRIAL: NCT00684333
Title: Assessment of Safety and Efficacy of EZ-Ject Injector a Novel Device for Pain-Free Subcutaneous Automatic Injection in Healthy Volunteers
Brief Title: Safety and Efficacy of EZ-Ject Injector a Pain-Free Subcutaneous Automatic Injection in Healthy Volunteers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Sindolor (Industry)
Responsible Party: Dr. Hanna Levy, Sindolor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: TRC 015/10062
Record Dates: First submitted 2008-05-19; First posted 2008-05-26 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: painless Injections; Subcutaneous Injections; Subcutaneous Injections to healthy volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- group 1 (Experimental): volunteers
  Interventions: Device: painless subcutaneous injection by EZ-Ject Injector

INTERVENTIONS:
Device: painless subcutaneous injection by EZ-Ject Injector — EZ-Ject Injector device employee cutaneous local anesthesia on the injection site by an electronic anesthetic system

SUMMARY:
Subcutaneous injections are a widely used method for drug delivery. One of its major drawbacks is the pain inflicted during the process. Sindolor has developed the chemical-free EZ-Ject Injector device, based on employing cutaneous local anesthesia on the injection site by an electronic anesthetic system. The purpose of this study is to determine the safety and efficacy of the EZ-Ject for subcutaneous injections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males and females between 18 and 50 years of age.
* Colour of skin that will enable to clearly observe dermal effects.
* Non-pregnant, non-lactating female subjects whose urine screening pregnancy test is negative.
* Subjects must be available to complete the study.
* Subjects must satisfy a medical examiner about their fitness to participate in the study.
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* Persons with a large amount of hair on the injection sites
* Presence of tattoos, discoloration, acne, scars, keloids or any other marks, bruises cuts or abrasions that could interfere with the observation of the injection sites.
* History of skin allergy or hypersensitivity
* History of severe skin infection in the past 1 year.
* History of easy bruising.
* Current or previous history of neurological disorders (particularly neuropathies), low back pain with neurological involvement.
* Any psychological condition that could influence the conduct of the study or interpretation of results.
* A history of drug or alcohol abuse
* Use of alcohol or medications within 48 hours prior to and during study participation
* Any condition, which in the opinion of the Principal Investigator or the study physician would place the subject at risk or influence the conduct of the study or interpretation of results.
* Inability to communicate well with the investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Study primary goal is to evaluate the safety of using the EZ-Ject Injector device for subcutaneous injections.The safety of using the EZ-Ject Injector device will be established by paucity of major complications that are device-related. | immediately

SECONDARY OUTCOMES:
Study secondary goal is to asses the efficacy of using the EZ-Ject Injector device. Efficacy will be assessed by alleviating injection pain. Subjective discomfort and pain will be assessed by analogue pain scale (VAS Scale). | immediately

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, M.D., Principal Investigator — Ichilov Medical center
Locations (1):
- Ichilov Medical center, Tel Aviv, Israel